CLINICAL TRIAL: NCT02959762
Title: Vitamin K to Slow Progression of Dyslipidemia and Diabetes Risk
Brief Title: Vitamin K to Slow Progression of Dyslipidemia and Diabetes Risk (Vita-K 'n' Kids Study II)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Norman Pollock, Associate Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 931430; 16GRNT31090037 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2016-10-11; First posted 2016-11-09 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Insulin Resistance; Obesity in Diabetes; Nutritional and Metabolic Diseases; Hyperlipidemia; Hyperglycemia; Cardiovascular Diseases
Keywords: G01 [Biological Sciences]; G02.513 [Nutrition]; G06.696.259 [Child Nutrition]; G07.553.481.398.571 [Obesity]; G06 [Biochemical Phenomena, Metabolism, and Nutrition]; G12.392.617 [Insulin Resistance]; G06.696.259.500 [Adolescent Nutrition]; A06 [Endocrine System]; A07 [Cardiovascular System]; C18.452.297.681 [Obesity in Diabetes]; C18.452.555 [Insulin Resistance]; C18 [Nutritional and Metabolic Diseases]; C18.452.494 [Hyperlipidemia]; C18.452.460 [Hyperglycemia]; C14 [Cardiovascular Diseases]; D11.786.875.844 [Vitamin K 2]; D02.806.550.750 [Vitamin K 2]; E02.293 [Diet Therapy]; E02 [Therapeutics]; F04.096.544.215.508.428 [Primary Prevention]; N01.224.425.525 [Nutritional Status]
MeSH Terms: conditions — Obesity; Insulin Resistance; Nutritional and Metabolic Diseases; Hyperlipidemias; Hyperglycemia; Cardiovascular Diseases; Metabolic Diseases | interventions — Vitamin K 2; menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo-Control (Placebo Comparator): The placebo-control group will take two placebo softgel capsules every day for 8 weeks.
  Interventions: Dietary Supplement: Placebo-Control
- Low-Dose Vitamin K2 (45-mcg/d) (Active Comparator): The low-dose vitamin K2 group will take one 45-mcg vitamin K2 softgel capsule and one placebo softgel capsule every day for 8 weeks.
  Interventions: Dietary Supplement: Low-Dose Vitamin K2 (menaquinone-7; 45-mcg/d)
- High-Dose Vitamin K2 (90-mcg/d) (Active Comparator): The high-dose vitamin K2 group will take two 45-mcg vitamin K2 softgel capsules every day for 8 weeks.
  Interventions: Dietary Supplement: High-Dose Vitamin K2 (menaquinone-7; 90 mcg/d)

INTERVENTIONS:
Dietary Supplement: Placebo-Control — two placebo softgel capsules per day (for 8 weeks) containing no vitamin K2 (menaquinone-7)
  Arms: Placebo-Control
Dietary Supplement: Low-Dose Vitamin K2 (menaquinone-7; 45-mcg/d) — one 45-mcg vitamin K2 (menaquinone-7) softgel capsule per day and one placebo softgel per day (containing no menaquinone-7) for 8 weeks
  Other Names: menaquinone-7
  Arms: Low-Dose Vitamin K2 (45-mcg/d)
Dietary Supplement: High-Dose Vitamin K2 (menaquinone-7; 90 mcg/d) — two 45-mcg vitamin K2 (menaquinone-7) softgel capsules per day for 8 weeks
  Other Names: menaquinone-7
  Arms: High-Dose Vitamin K2 (90-mcg/d)

SUMMARY:
Animal studies have found that vitamin K-dependent proteins matrix Gla protein and osteocalcin beneficially influence lipid and glucose metabolism, respectively. However, this concept has not been tested in humans at risk for dyslipidemia and diabetes risk. Vitamin K supplementation presents an opportunity to test the hypothesized link between the vitamin K-dependent proteins and markers of lipid and glucose metabolism. The investigators will conduct an 8-week vitamin K intervention (to manipulate carboxylation of matrix Gla protein and osteocalcin) and determine its effects on markers of dyslipidemia and diabetes risk. Sixty obese children will be randomly allocated to either the control group receiving placebo or the low-dose (45 mcg/d) or high-dose group (90 mcg/d) receiving vitamin K (menaquinone-7).

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 17 years
* Body mass index equal to or greater than 85th percentile for age and sex
* Subject and parent/guardian understands the study protocol and agrees to comply with it
* Informed Consent Form signed by the parent/guardian and assent signed by the subject

Exclusion Criteria:

* Subjects using vitamin supplements containing vitamin k
* Subjects with (a history of) metabolic or gastrointestinal diseases including hepatic disorders
* Subjects presenting chronic degenerative and/or inflammatory diseases
* Subjects receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters (salicylates, antibiotics)
* Subjects receiving corticosteroid treatment
* Subjects using oral anticoagulants
* Subjects with a history of soy allergy
* Subjects who have participated in a clinical study more recently than one month before the current study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum lipid concentrations | 8 weeks
  To determine if the vitamin K-induced change in matrix Gla protein carboxylation improves fasting lipid panel (triglycerides, total cholesterol, HDL-cholesterol, and LDL-cholesterol) in a dose-dependent manner.
Change in insulin sensitivity | 8 weeks
  To determine if the vitamin K-induced change in osteocalcin carboxylation effects insulin sensitivity in a dose-dependent manner. Insulin sensitivity will be calculated from plasma insulin and glucose concentrations measured during a two-hour oral glucose tolerance test by using the oral glucose minimal model.
Change in beta-cell function | 8-weeks
  To determine if the vitamin K-induced change in osteocalcin carboxylation effects beta-cell function in a dose-dependent manner. Beta-cell function, as assessed by dynamic beta-cell responsitivity, will be calculated from plasma glucose and C-peptide concentrations measured during a two-hour oral glucose tolerance test by using the oral C-peptide minimal model.

SECONDARY OUTCOMES:
Change in coagulation | 8 weeks
  Coagulation-related parameters (i.e., prothrombin time and activated partial thromboplastin time) will be assessed at baseline and 8 weeks to assess clotting function.
Change in arterial stiffness (pulse wave velocity) | 8 weeks
  Arterial stiffness, as measured by pulse wave velocity (PWV), will be assessed at baseline and 8 weeks to explore whether change in arterial stiffness is influenced by vitamin K2 supplementation.
Change in endothelial function (flow-mediated dilation) | 8 weeks
  Endothelial function, as measured by flow-mediated dilation (FMD), will be assessed at baseline and 8 weeks to explore whether change in endothelial function is influenced by vitamin K2 supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Pollock, PhD, Principal Investigator — Department of Pediatrics, Medical College of Georgia, Augusta University
Locations (1):
- Medical College of Georgia; Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
1. Approximate date of when the data will be shared? 2019-06-28
  2. Where will the data be made available? The de-identified data will be made available for research purposes only by contacting the principal investigator.
  3. Please explain any limits to data sharing that might be required. Even though the final research data will be stripped of identifiers prior to release for sharing, the investigators believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, the investigators will make the data available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Douthit MK, Fain ME, Nguyen JT, Williams CF, Jasti AH, Gutin B, Pollock NK. Phylloquinone Intake Is Associated with Cardiac Structure and Function in Adolescents. J Nutr. 2017 Oct 1;147(10):1960-1967. doi: 10.3945/jn.117.253666. PMID 28794209